CLINICAL TRIAL: NCT06962202
Title: Modified Desmopressin (Mdesmo Cold-Kit) for PET Imaging to Localize Adrenocorticotropic Hormone (ACTH) Dependent Cushing Syndrome (CS)
Brief Title: Modified Desmopressin (mDesmo) Using Cold-Kit for PET/CT
Acronym: Ga-68 mDesmo
Status: Recruiting | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, Jaya Shukla, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: PGI/IEC/2021/001537; TDP/BDTD/59/2021(G) (Other Grant/Funding Number: Department of Science and Technology, New delhi India); CTRI/2022/08/044615 (Registry Identifier: Clinical Trials Registry-India)
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cushing Syndrome
Keywords: ACTH; bilateral inferior petrosal sinus sampling; Corticotropinoma; transsphenoidal surgery; PET/CT
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Surgical samples for histopathological examination fpr correlation with imaging data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cushing syndrome (CS) characterized by excessive cortisol secretion in the body: To detect and localize the tumor responsible for ACTH-dependent CS. For deleneation of small tumors within the pituitary. Ga-68mDesmo will be injected to enable PET/CT imaging. Ga-68 is a positron emitter.

SUMMARY:
The incidence of Cushing syndrome (CS) is 1.2-3.2 cases per million per year, of which adrenocorticotropic Hormone (ACTH)-dependent disease comprises approximately 70-80% of cases. Among these, nearly 90% of ACTH-dependent CS are due to pituitary-dependent CS, known as Cushing disease (CD). The management of ACTH-dependent CS relies on distinguishing Cushing disease (or Corticotropinoma) from ectopic Cushing syndrome (ECS) followed by localization of the tumor in the sella. The diagnosis of CD is very challenging, especially when they are microadenomas (<6 mm). Current imaging techniques, such as magnetic resonance imaging (MRI), have limitations in accurately delineating (sensitivity 60%) these tumors. Even if the lesion is detected inside the pituitary, the functionality of the tumor is questionable, as there can be innocent pituitary tumors which actually are not the cause of Cushing syndrome in a particular case. The diagnosis gets more complex with the fact that 10% of the ECS cases are reported to have an incidental non-functioning pituitary tumor, this can complicate the diagnosis of ECS. Though the localizing accuracy of bilateral inferior petrosal sinus sampling (BIPSS) is 90%, the lateralization (40-70%) of corticotropinoma (whether the lesion is located on the right or left side) based on BIPSS is still questionable. These challenges contribute to the fact that in approximately 30% of cases of CD, the source of ACTH excess remains occult. The lack of information on accurate localization and lateralization of corticotropinoma leads to reduced remission rates after surgery. Therefore, novel approaches to diagnosing Cushing disease are needed.

We have developed a novel radiopharmaceutical Gallium-68- 1,4,7,10-tetraazacyclododecane-N,N',N',N'-tetraacetic acid-modified desmopressin (68Ga-DOTA-mDesmo) for Positron Emission Tomography/Computed Tomography (PET/CT). This radiopharmaceutical has the potential to selectively target the overexpressed V1b receptors in patients diagnosed with Cushing disease. The clinical studies demonstrated 100% diagnostic accuracy of 68Ga-DOTA-mDesmo PET/CT in delineating corticotropinomas, surpassing the accuracy of CE-MRI and BIPSS, regardless of adenoma size. However, the small sample size and regional patient recruitment may affect the generalizability of the results.

The project aims to assess the diagnostic sensitivity and specificity of 68Ga-DOTA-mDesmo in a diverse Cushing syndrome population. This will lead to development and validation of a superior, non-invasive diagnostic modality for accurate corticotropinoma delineation, aiding neuro-navigation during surgery and potentially improving treatment outcomes for ACTH-dependent Cushing syndrome.

DETAILED DESCRIPTION:
Cushing's syndrome (CS) is one of the most enigmatic endocrine disorders. It is important to confirm the adrenocorticotropic Hormone (ACTH) dependent hypercortisolism and distinguishing Cushing's disease from ectopic CS. Most of the ACTH dependent CS are caused by Cushing's disease, of which majority are due to microadenoma being less than 6 mm. Visualizing tumors within 10 mm pituitary and confirming its functional status is challenging. Long-term remission/cure is determined by the correct functional and anatomical delineation of corticotropinoma (pituitary-tumor). The treatment of choice in Cushing's disease is pituitary microsurgery also known as transsphenoidal surgery (TSS). However, pituitary-tumor is not well delineated within the sella in 30-40% using currently available investigations especially MRI and inferior petrosal sinus sampling, which affects intra-operative navigation for selective adenectomy and influence remission rate. The modified Desmopressin (mDesmo) was synthesized to be conjugated with 1,4,7,10-tetraazacyclododecane-N,N',N',N'-tetraacetic acid (DOTA) and radiolabelled with Gallium-68 (Ga-68), a positron emitter, for Positron Emission Tomography/Computed Tomography (PET/CT) imaging to delineate pituitary-tumor. It provides surgeon with the requisite information for intra-operative tumor navigation.

Objectives of the Project

1. Preparation of freeze-dried DOTA conjugated mDesmo cold-kit for radiolabelling with Ga-68 and PET/CT imaging.
2. Bioevaluation of radiotracer prepared with mDesmo cold-kit for the molecular imaging of ACTH-releasing pituitary adenoma (Cushing's disease).
3. Evaluate the application of Ga-68 mDesmo PET/CT in intra-operative tumor navigation, residual disease and recurrence.
4. Study the self-life of mDesmo cold-kit.

Deliverables:

Cushing's syndrome may be due to a) extra pituitary tumors (also known as EAS or ECS) that can be easily detected by Gallium-68-1,4,7,10-tetraazacyclododecane-N,N',N',N'-tetraacetic acid Tyr3-octreotate/Nal3-octreotide (68GaDOTATATE/NOC) and resected, b) tumors within the pituitary (known as pituitary corticotropinoma). Many a times these tumors are very small (<6mm, microadenoma). The treatment of choice is pituitary microsurgery (trans-sphenoidal surgery). However, the correct delineation of these microadenomas within small pituitary (10 mm) before microsurgery is challenging but crucial to preserve normal functioning pituitary.

None of the currently available diagnostic modalities can delineate the tumor from normal functional pituitary. Often MRI and BIPSS, an invasive and overly expensive, is used to guide surgery.

Therefore

* The mDesmo cold-kit has been developed for PET/CT imaging as single modality to correctly delineate microadenomas noninvasively.
* Provides surgeon with the requisite information for intra-operative tumor navigation
* Cost-effective
* Facile procedure of radiolabelling
* Developed first time globally
* International market Significance of the Project

  1. Major applications of the proposed technology Cushing's syndrome (CS) is a rare endocrine disorder. The diagnosis can be challenging due to the non-specific nature of many symptoms. On suspicion of the disease, it is important to confirm the presence of ACTH dependent hypercortisolism. Seventy to 80% cases of ACTH dependent Cushing's syndrome are caused by Cushing's disease (pituitary tumor), of which 90% are due to microadenoma of less than 6 mm. Visualizing these small tumors within 10 mm pituitary and confirming its functional status is a challenge. In patients with clinically and biochemically confirmed endogenous Cushing's syndrome, the long-term remission/cure is determined by the correct functional and anatomical delineation of corticotropinoma (pituitary tumor) i.e. to distinguish between Cushing's disease (access ACTH production within pituitary due to tumor) and ectopic ACTH production (Corticotrophin-releasing hormone (CRH) producing tumors outside pituitary) and most importantly, correct visualization of tumour, preoperative. The ectopic ACTH syndrome require resection of the primary tumour while the treatment of choice in Cushing's disease is pituitary microsurgery. Corticotropinoma is not well delineated within the sella in 30 to 40% cases of Cushing's disease using currently available investigations especially MRI and bilateral inferior petrosal sinus sampling (BIPSS), which affects intra-operative navigation for selective adenomectomy and thus may influence remission rates after trans-sphenoidal surgery (TSS).

     Anatomical imaging (Computed Tomography (CT), Magnetic Resonance Imaging (MRI) can delineate the tumor while cannot confirm its functionality, while vice versa is true for functional test/imaging. None of the currently available diagnostic modality can achieve these goals simultaneously. Several tests are used to serve this purpose. However, none of the tests are diagnostic. Pituitary tumor i.e corticotropinoma continues to express receptors for Corticotropin releasing hormone (CRH) and Arginine vasopressin (AVP) as that of normal corticotrophs and rather corticotropinoma hyper responds to these stimuli due to upregulation of the respective receptors.

     Desmopressin, a small peptide consist of 9 amino acids, is more potent and specific for tumorous corticotrophs, therefore we explored this molecule for PET/CT imaging. The native Desmopressin could not be conjugated to bifunctional chelator for radionuclide binding, some modifications were done in amino acid sequence of Desmopressin to conjugate with bifunctional chelator (DOTA in this case) without affecting it binding property with receptor. The modified and DOTA conjugated desmopressin (mDesmo) when radiolabelled with Gallium-68 (Ga-68 mDesmo), the PET/CT hybrid imaging is able to delineate cortitropinoma i.e. integrated functional imaging of tumor with anatomical localization and provides surgeon with the requisite information for intra-operative tumor navigation.
  2. Clinical Need (Include significance and estimated patient population/year if known).

Cushing's syndrome is a clinical state resulting from inappropriate and excess production of cortisol. This syndrome may arise due to excessive adrenocorticotrophic hormone (ACTH) production from the pituitary gland or ACTH/ corticotropin releasing hormone (CRH) secretion from an extra-pituitary source or autonomous cortisol secretion from adrenal glands. The incidence of Cushing's syndrome is 1·2-2·4 cases per million per year, of which 80% is due to excess ACTH production (1). Amongst the ACTH dependent causes, Cushing's disease is the most common cause seen in 90% of cases, the rest being due to ectopic ACTH/CRH production (ECS). In most of the cases, Cushing's disease is caused by micro-corticotropinoma of less than 6 mm (2). The localization the source of ACTH is crucial for management. This begins with Contrast enhanced Magnetic resonance imaging (CEMRI) of sella as Cushing's disease constitutes 90% of ACTH dependent Cushing's syndrome (3). However, CEMRI has a sensitivity of 50 to 60% with a positive predictive value of 86% (2). Furthermore, it is an anatomical imaging and do not indicate the functional status of the tumor. It may reveal innocent pituitary incidentaloma in up to 10% of the general population including patients with ectopic Cushing's syndrome (ECS) (4). Thereby, meaning that these pituitary tumor picked up on MRI may just be an incidental finding and not the actual culprit behind the symptomatology. While the presence of macroadenoma favours pituitary source of ACTH, the presence of microadenoma warrants further corroboration with the functional/dynamic tests for the confirmation of corticotropinoma which include high dose dexamethasone suppression test (HDDST), CRH stimulation test and bilateral inferior petrosal sinus sampling (BIPSS). The pre- test probability of having pituitary disease in ACTH dependent CS is between 85 to 90%, which makes it mandatory for any additional dynamic test to be of any clinical use to have a high specificity. Patients with concordant response to CRH stimulation and HDDST indicating pituitary source are almost certain to harbour corticotropinoma. However, in case of discordant results and/or non-yielding MRI, BIPSS is required (5). Importantly, BIPSS is an invasive procedure which is limited by its availability, need for high degree of technical skill and cost. Even though it is a good modality for differentiating ectopic from pituitary source of ACTH production, its positive predictive value for corticotropinoma lateralization within pituitary as indicated by inter sinus ACTH ratio is only 60-70% (5). Furthermore, it does not provide sufficient information for planning surgical navigation, due to which surgeries solely based on lateralization as indicated by inter-sinus ACTH gradient on BIPSS leads to only 45% cure rates (6). Thus, with the current modalities, corticotropinoma is not well delineated within the sella in 30 to 40% cases of Cushing's disease. This affects intra-operative navigation for selective adenomectomy which may influence remission rates after trans-sphenoidal surgery (TSS).

Currently there is no imaging modality available globally that can give functional and anatomical details of ACTH dependent pituitary adenoma. Earlier we have developed Ga-68 CRH for this purpose and evaluated clinically in patients with ACTH dependent Cushing's Syndrome (8). However, being a large peptide of 41 amino acid there was high uptake of Ga-68 CRH in liver. it also demonstrated diffuse physiological uptake in normal pituitary and other organs (9).

Desmopressin is deamino D-arginine vasopressin (DDAVP) is found more potent and specific than arginine vasopressin (AVP) and CRH for tumorous corticotrophs. Therefore, we explored this molecule for PET/CT imaging of ACTH dependent pituitary adenoma. Desmopressin was modified to enable radiolabelling with PET radionuclide Ga-68. Ga-68 mDesmo PET/CT provide functional as well as anatomical information to delineate corticotropinoma, provide surgeon with the requisite information for intra-operative tumor navigation and preservation of normal pituitary.

The aim of the study is to develop a non-radioactive (cold kit) formulation. so that the same may be available to all hospital based radiopharmacy for quick and a facile synthesis of PET tracer, Ga-68 mDesmo, for lateralizing pituitary adenoma (Cushing's disease) and differential diagnosis of ACTH-releasing pituitary adenoma (Cushing's disease) from the of ectopic ACTH-secreting tumors by non-invasive molecular imaging (PET/CT).

References

1. Loriaux DL. Diagnosis and Differential Diagnosis of Cushing's Syndrome. Longo DL, editor. N Engl J Med. 2017 Apr 13;376(15):1451-9.
2. Aron DC, Raff H, Findling JW. Effectiveness Versus Efficacy: The Limited Value in Clinical Practice of High Dose Dexamethasone Suppression Testing in the Differential Diagnosis of Adrenocorticotropin-Dependent Cushing's Syndrome. J Clin Endocrinol Metab. 1997 Jun 1;82(6):1780-5.
3. Jarial KDS, Bhansali A, Gupta V, Singh P, Mukherjee KK, Sharma A, et al. Diagnostic accuracy and comparison of BBIPSS in response to lysine vasopressin and hCRH. Endocr Connect. 2018 Mar;7(3):425-32.
4. Oldfield EH, Doppman JL, Nieman LK, Chrousos GP, Miller DL, Katz DA, et al. Petrosal Sinus Sampling with and without Corticotropin-Releasing Hormone for the Differential Diagnosis of Cushing's Syndrome. N Engl J Med. 1991 Sep 26;325(13):897-905.
5. Dickstein G, DeBold CR, Gaitan D, DeCherney GS, Jackson RV, Sheldon WR, et al. Plasma corticotropin and cortisol responses to ovine corticotropin-releasing hormone (CRH), arginine vasopressin (AVP), CRH plus AVP, and CRH plus metyrapone in patients with Cushing's disease. J Clin Endocrinol Metab. 1996 Aug;81(8):2934-41.
6. Cassarino MF, Sesta A, Pagliardini L, Losa M, Lasio G, Cavagnini F, et al. Proopiomelanocortin, glucocorticoid, and CRH receptor expression in human ACTH-secreting pituitary adenomas. Endocrine. 2017 Mar;55(3):853-60.
7. Boyle, J., Patronas, N.J., Smirniotopoulos, J. et al. CRH stimulation improves 18F-FDG-PET detectionof pituitary adenomas in Cushing's disease Endocrine (2019) 65: 155
8. Walia R, Gupta R, Bhansali A, ........ Shukla J. Molecular Imaging Targeting Corticotropin Releasing Hormone Receptor for Corticotropinoma: A Changing Paradigm. J Clin Endocrinol Metab. 2020 Oct 20:dgaa755.
9. Shukla J Vatsa R, Chhabra R, Rana N, Kumar R, Singh H, Mittal BR, Walia R. Development of DOTA conjugated synthetic Corticotrophin Releasing Hormone (CRH) for PET/CT imaging of ACTH Dependent Cushing's Disease. accepted. Cancer Biother Radiotherapy 2021.

10 Nieman LK, Biller BMK, Findling JW, Newell-Price J, Savage MO, Stewart PM, et al. The Diagnosis of Cushing's Syndrome: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2008 May 1;93(5):1526-40.

STATUS OF DEVICE IDEA The product mDesmo has been custom synthesized and radiolabelled with high labelling efficincy. The clinical studies were also performed after obtaining clearance from Institutional Ethics Committee.

Ga-68 mDesmo is found promising agent for delineation of corticotropinoma and intra-operative navigation. Since Ga-68 has half-life of only 68 min, the proposed solution for application is to prepare a cold kit (non-radioactive formulation) that can be used after radiolabelling at any hospital/Center having PET/CT scanner. This may be a breakthrough in the pituitary microadenoma. it may pinpoint the tumor (delineate) for remission surgery and preserve the pituitary.

Structural modification of ligand molecule Desmopressin is a 9 amino acids peptide, and we have modified the structure for the suitability of conjugation of bifunctional chelating agent for radiolabeling and receptor binding affinity. The current molecule is a 10 amino acid peptide. We have given the name modified desmopressin or mDesmo.

Radiolabelling and quality control Our experimental data demonstrates >99% radiolabeling yield and radiochemical purity of 68Ga-mDesmo. The quality control tests of in-house synthesized 68Ga-mDesmo such as shelf-life, stability, sterility, and pyrogenicity tests indicate the suitability of radiotracer for intravenous administration.

Shelf-life and Stability Shelf-life of the in-house synthesized 68Ga-mDesmo was assessed in saline at room temperature for 4 hours. Similarly, stability was assessed in PBS and in human-serum at 37oC for 4 hours. The prepared radiopharmaceutical was found to be stable for up to 4 hours with a shelf-life of 4 hours.

Sterility For sterility assessment, 1 mL of 68Ga-mDesmo was incubated separately in 10 mL fluid thioglycollate medium (FTM) and 10 mL tryptic soy broth (TSB). The FTM culture was incubated at 25oC for 14 days and TSB culture was incubated at 35oC for 14 days. Negative control of both media was also incubated. The cultures were monitored on daily basis for turbidity. The preparation was found to be free from any microbial contamination as no visible growth or turbidity was observed up to 14 days in both mediums.

Pyrogenicity The end-point chromogenic Limulus Amebocyte Lysate (LAL) test was performed to assure the absence of unsafe levels of bacterial endotoxin pyrogen in radiopharmaceutical preparation. The specification value of endotoxins in the preparation for intravenous administration is not more than 175 Endotoxin Unit (EU)/V, where V is the volume of injection. The endotoxin value of 68Ga-mDesmo injection was found to be 7.5 EU/V, which was well within the range, and the preparation was considered for intravenous administration.

Clinical Study Pilot clinical studies were performed after obtaining clearance from Institutional Ethics Committee (IEC-08/2019-1353, dated 22 October 2019). Informed consent was also obtained from the patients. There was no physiological uptake of Ga-68 mDesmo observed throughout in body including normal pituitary. Visualization of kidney and bladder indicate the renal route of excretion of Ga-68 mDesmo. High blood pool activity was also observed at 1h and 2 h. Good tumor to background ratio in patients indicated the diagnostic potential of 68Ga-mDesmo for delineating Cushing's disease from ectopic ACTH secreting tumors.

CURRENT CLINICAL PRACTICES None of the currently available diagnostic modality can achieve these goals simultaneously. Therefore, a battery of tests is used to serve this purpose and described below. However, none of the tests are diagnostic.

Assessment of clinical symptoms Cushing's syndrome is a clinical condition characterized by excessive circulating cortisol and by various clinical features such as gain of weight, menstrual, disturbances, hirsutism, psychiatric dysfunction, proximal muscle weakness, osteoporosis, fractures, loss of scalp hair, plethora, rounding of face, hypertension, easy bruising, wide purple striae, (>1cm) hyper pigmentation, and diabetes.

History of Medication Cushing syndrome can be due to exogenous or endogenous causes. Exogenous Cushing's syndrome occurs due to excessive use of glucocorticoids whereas endogenous Cushing's syndrome is induced by inappropriate secretion of cortisol owing to abnormalities in the hypothalamic pituitary adrenal (HPA) axis. The anterior pituitary gland leading to release of adrenocorticotropic hormone (ACTH). Further, ACTH binds to receptors present on the adrenal cortex and stimulates the release of cortisol. Excessive production of ACTH from the pituitary gland or from ectopic source (non-pituitary) triggers the excessive release of cortisol from adrenals resulting in Cushing's syndrome. Pituitary microsurgery is one of the major tools to cure the Cushing's disease, for this an accurate localization of the tumor, to preserve normal pituitary functions, is essential requirements.

Biochemical Tests Cortisol dynamics included 08:00 and 23:00 hour cortisol and ACTH, overnight dexamethasone suppression test (ONDST), low dose dexamethasone suppression test (LDDST) and high dose dexamethasone suppression test (HDDST) as per standard protocol.

Imaging Pre-operative imaging of the pituitary by contrast-enhanced Magnetic Resonance Imaging and this technique has a sensitivity of 70%. Pituitary tumors were divided into not-visualized (NV), microadenoma (<10 mm) and macroadenoma (≥10 mm). In patients with non-visualized pituitary tumor or suspicion of Ectopic Adrenocorticotrophin (ACTH) secretion (EAS), CT neck, thorax and abdomen and somatostatin receptor-based scintigraphy is performed.

Anatomical imaging (CT, MRI) can delineate the tumor while cannot confirm its functionality, while vice versa is true for functional test/imaging. Pituitary tumor i.e corticotropinoma continues to express receptors for Corticotropin releasing hormone (CRH) and Arginine vasopressin (AVP) as that of normal corticotrophs and rather corticotropinoma hyper responds to these stimuli due to upregulation of the respective receptors.

Gold Standard Bilateral inferior petrosal sinus sampling (BIPSS) is an invasive, technically demanding test with limited availability due to high cost, globally. Intravenous administration of CRH/desmopressin is used during BIPSS to stimulate ACTH production. It has sensitivity and specificity of more than 95% for differentiation of pituitary vs. ectopic production of ACTH. However, lateralization accuracy that is the ability to lateralize the side of corticotropinoma in the pituitary is only 70%, thereby limiting its utility to guide surgical procedure. Surgery done based on BIPSS results in cure rate of 50-60%. BIPSS has been associated with comorbid and even fatal complications, including deep venous thrombosis, pulmonary emboli, and brain stem vascular damage. Since the procedure is technical and invasive, experienced teams will have better results and fewer complications. CRH used in BIPSS is generally safe but may be associated with mild side effects like tachycardia, hypotension, dizziness and flushing. However, it is very expensive.

Vasopressin though causes several side effects such as abdominal pain or cramps, nausea, vomiting, pale skin, increased urge to bowl movements, dizziness, light headedness and hypertension but relatively cost-effective.

Other Molecular Imaging One study used Fluorodeoxyglucose-18 (FDG) PET/CT after intravenous cold CRH and suggested that giving CRH prior to PET improved its efficacy for detecting pituitary tumor. However, FDG is a nonspecific agent and the uptake of this is dependent on the metabolic activity of the tumour and is taken up by all other pituitary tumours. More-over, the interpretation of FDG PET/CT is difficult as even brain parenchyma has a bright uptake of FDG.

Our group had also developed Ga-68 CRH to image ACTH dependent Cushing's syndrome and the patient's data is published. Ga-68 CRH is a promising agent to delineate corticotropinoma and intra-operative navigation. Ga-68 CRH is the only competitor molecule of our proposed molecule (Ga-68 mDesmo).

SUPERIORITY OF DEVICE AS COMPARED TO EXISTING DEVICES AND PRACTICES Cushing disease is the commonest cause of ACTH-dependent Cushing's syndrome (90%). Transsphenoidal surgery is the treatment of choice. However, a battery of tests are required to confirm the disease, rule out associated conditions and delineate (pinpoint) the tumor that needs to be removed. As described above BIPSS is invasive, expensive and require specialized (skilled) person to perform the procedure. Additionally, all these tests have limited sensitivity and specificity.

We have also developed Ga-68 mDesmo which can be used as non-invasive imaging technique to pinpoint functional tumor. In our clinical studies, it is found suitable for delineating corticotropinoma and intra-operative navigation. Most importantly, there was no physiological uptake of Ga-68 mDesmo throughout in body including normal pituitary. Visualization of kidney and bladder indicate the renal route of excretion of Ga-68 mDesmo (Fig 1).

The promising results inspired us to think for a formulation that can be commercially available for radiolabelling and PET/CT imaging. The Ga-68 is half-lived life of only 68 mins. Therefore, non-radioactive freeze-dried formulation with facile radiolabeling protocol for hospital based radiopharmacy would be the most suited and ideal option. As no such molecule is currently available globally, this ready to use formulation seems very promising. 68Ga-mDesmo PET/CT imaging will delineate the corticotropinoma from EAS without further performing invasive and costly test like BIPSS. It will also provide surgeons the requisite information for intra-operative tumor navigation.

REVIEW OF STATUS AND TECHNOLOGY TRENDS IN RESPECT OF DEVICE TO BE TAKEN UP FOR DEVELOPMENT:

1. Patients of Cushing's syndrome can be treated based on etiology of tumors. i. Cushing's Disease-Transsphenoidal surgery (CD/TSS) - Disease remission ii. Cushing's Disease-Total bilateral adrenalectomy (CD/TBA) for symptomatic relief iii. Ectopic Adrenocorticotrophin (ACTH) secretion (EAS)-removal of primary tumor
2. Based on size, the pituitary tumors may be divided non-visualized (NV), micro- and macroadenoma. Macroadenomas are well characterized on CEMRI. However, the challenge lies on the pinpointing the microadenoma and non-visualized.
3. Though ACTH correlates with the tumor size, but it is very challenging to differentiate micro-and macroadenoma on clinico-biochemical basis.
4. CEMRI represents a pure anatomical imaging and limited by its poor sensitivity and inability to differentiate between functioning adenoma and pituitary incidentalomas.
5. The current guidelines recommend BIPSS in cases of ACTH dependent CS where adenoma size is less than 6 mm or dynamic testing shows discordant results (10). However, factors that limit its use are lack of widespread availability, need for high degree of technical expertise, cost and potential adverse events due to it being an invasive procedure. Therefore, very limited number of patients could undergo BIPSS. Moreover, BIPSS is mainly meant for localizing the source of excess ACTH to either pituitary or extra-pituitary site. The low positive predictive value for lateralization (40-70%), leads to limited benefit in post-surgical remission rate (45%). BIPSS does not have any role in Cushing's disease recurrence and being invasive.

18F-FDG and 11C-methionine PET-CT have been used to delineate corticotropinoma with a limited success as these are non-specific imaging based on glucose metabolic and protein synthesis.

These limitations may easily be overcome by non-invasive 68Ga-mDesmo PET-CT imaging. The physiological uptake is not seen in normal pituitary. The 68Ga-mDesmo PET-CT is based on of binding of 68Ga-mDesmo to V3 receptors on corticotropinoma that are absent on normal pituitary as observed in imaging.

As compared to other nuclear imaging modalities, 68Ga-mDesmo PET/CT:

i) is more sensitive and provide functional status of tumor; ii) functional and anatomical fused images are more suitable for localization of corticotropinoma for conservation surgery; iii) To evaluate surgical therapy and information of residual tumor; iv) information of recurrent tumor for management (gamma-knife vs surgical resection).

The promising results of 68Ga-mDesmo PET/CT imaging inspired us to think for a formulation that can be commercially available for solving the most challenging situation regarding the most important gland of the human body.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with endogenous Cushing's syndrome
2. Patients in the age group of 5 to 75 years.
3. Patients willing to give informed consent.

Exclusion Criteria:

1. Patient with exogenous exposure to steroids
2. Ongoing pregnancy
3. Severe comorbid conditions that may interfere with the study.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 100 Pts with Cushing Syndrome and 5 control patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
PET/CT Imaging with Ga-68mDesmo | one day
  Precise localization of corticotropinoma (ACTH secreting tiny adenoma in pituitary)

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Sciences, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
currently it is a single centric study, therefore, it will not be ethical to share data with other researchers.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-05-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT06962202/Prot_SAP_ICF_000.pdf